CLINICAL TRIAL: NCT04644263
Title: Turkish Validity and Reliability of The Tampa Scale for Kinesiophobia for Temporomandibular Disorders
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Eylem KÜÇÜK, Head of Physiotherapy, Okan University
Other Study IDs: Eylem Kucuk, OkanU
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validity and reliability

SUMMARY:
Objective: The aim of this study is to evaluate the validity and reliability of the Turkish version of the 'The Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-TMD)' questionnaire used to assess kinesiophobia in temporomandibular joint disorders.

Method: The "Tampa Kinesiophobia Scale in Temporomandibular Disorders" (TSK-TMD), which consists of 12 item, was adapted to Turkish with the translation and back-translation method. 111 patients (75 females, 36 males) who had been diagnosed with temporomandibular joint for at least 6 months and diagnosed as Temporomandibular Joint Disorder were participated to fill out the questionnaire. In the present study, participants were assessed with the Temporomandibular joint disorders evaluation form, Turkish TSK-TMD-12 item, Visuel Analogue Scale (VAS) and Pain Catastrophizing Scale (PCS). The internal consistency and test-retest reliability with a 3-5 days time were used to evaluate the reliability of the TSK-TMD. The reliability of the corelatıon was checked with PCS. Construct validity was assessed based on conﬁrmatory factor analysis (CFA).

DETAILED DESCRIPTION:
We used Turkish TSK-TMD-12 item, Visuel Analogue Scale (VAS) and Pain Catastrophizing Scale (PCS) questionnaires in our study.

ELIGIBILITY:
Inclusion Criteria::

* volunteer participation in the study, between 18 and 65 years old,
* having symptoms for at least 6 months,
* being literate, and having communication to understand and answer questions.

Exclusion Criteria:

* toothache
* Cognitive impairment affecting their ability to understand and complete the study questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-test: 10 patients temporomandibular disorders evaluated. Inclusion and exlusion criteria listed above.
  Validation and reliability: 111 patients with temporomandibular disorders evaluated.Inclusion and exlusion criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
The Tampa Scale for Kinesiophobia for Temporomandibular Disorders | The measurement is one-time and take 20 minutes. It take an average of 6 month after the data of all participants are collected.
  The original TSK-TMD is an English scale and consists of 18 items to evaluate the fear of movement in TMD patients. 4-point Likert type scoring is used (1-strongly disagree, 2-partially disagree, 3-partially agree and 4- strongly agree). Total score is calculated by reversing 4, 8, 12, 16 items. In this short form, by collecting all points, scores between 12-48 are obtained. The higher the person's score indicates, the higher the kinesiophobia. They suggested that the 12-item version had good reliability and validity as a result of the structural reliability assessment and was more suitable for evaluation in TMD patients.
Pain Catastrophizing Scala | The measurement is one-time and take 15 minutes. It take an average of 6 month after the data of all participants are collected.
  It is a scale developed to detect catastrophic thoughts or feelings and ineffective coping methods of pain experienced by patients in the past. It describes the different thoughts and feelings that individuals can experience while suffering. PCS is a scale consisting of thirteen items and three factors such as helplessness, enlargement and self-reflection. Likert type scoring is evaluated between 0-4 points. The total score ranges from 0-52.